CLINICAL TRIAL: NCT00531258
Title: The Use of Non Invasive Brain Stimulation in the Treatment of the Sequelae of Closed Brain Injury
Brief Title: TMS in the Treatment of the Sequelae of Closed Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 011007
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Depression; Closed Head Injury
Keywords: Depression; TBI; TMS; Major Depression resulting from a mild to moderate closed head injury
MeSH Terms: conditions — Depression; Head Injuries, Closed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Device: rTMS
- 2 (Placebo Comparator)
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: rTMS — Bilateral rTMS
  Arms: 1
Device: Sham rTMS — sham rTMS
  Arms: 2

SUMMARY:
Depression is very common in people who have experienced a traumatic brain injury. Few treatments have been found to be effective in treating depression in this situation. We intend to investigate the effectiveness of a form of brain stimulation, transcranial magnetic stimulation, which has been found to be effective in treating depression in people who have not undergone a brain injury. By evaluating new methods of treating depression in this population, we hope to increase the options available for treating people in this difficult situation. Furthermore, problems with aspects of thinking are also commonly present post brain injury, as in some individuals with depression. Various brain stimulation techniques, including transcranial magnetic stimulation (TMS) have been shown to have a positive effect on cognition. We also intend to investigate whether a therapeutic effect on cognitive deficits is present following TMS, in addition to any effects on depression. New treatment protocols will be developed, and understanding of the pathology and treatment of post traumatic brain injury depression will be enhanced.

DETAILED DESCRIPTION:
It is plausible to propose that the same treatment paradigm may result in an improvement in mood and cognition with the possibility that these changes will be self reinforcing resulting in enhanced quality of life and reduced service demands.

The proposal for the use of rTMS in the treatment of post TBI depression is also supported by aetiological models. In particular, rTMS would seem to have considerable potential to improve pathophysiological changes relevant to the treatment of post TBI depression and cognitive dysfunction. Early models of the mechanism of action of rTMS treatment in depression were based on the observation that rTMS is able to produce localised changes in cortical activity [7]. The standard treatment paradigm generally has been found to produce an increase in local prefrontal cortical excitability. However, more recently there has been an increased understanding that rTMS modulates distal brain regions as well and potentially the strength of connections between brain regions. It has been proposed that its therapeutic effects in non TBI-related depression occur through modulation of dorsal frontal - subcortical limbic connectivity and potentially the actual integrity and strength of connections between these regions. If this is the case, altering cortical - cortical or cortical - subcortical connectivity may lead to therapeutic benefits in post TBI depression due to likely involvement of white matter changes in the development of TBI related mood disorder.

Aims/Objectives/Hypothesis/es Primary Aim: To assess the effectiveness of rTMS in treating depression post traumatic brain injury.

Secondary Aim: To gain preliminary data as to the possible effectiveness of rTMS in treating cognitive deficits post traumatic brain injury.

Hypothesis 1: Active bilateral sequential rTMS will lead to an improvement in the symptoms of post TBI depression, as measured by MADRS scores, when compared to sham treatment Hypothesis 2: Active bilateral sequential rTMS will lead to an improvement in cognitive executive functioning in individuals post TBI, when compared to sham treatment Hypothesis 3: Active bilateral sequential rTMS will lead to an improvement in life satisfaction and level of functioning in individuals post TBI, when compared to sham treatment.

Methodology Experimental Design and Randomisation Procedures The study has been designed to allow the reporting of results in a manner consistent with the international CONSORT guidelines. The study will involve a 4-week (20 session) randomized double-blind clinical trial with 2 treatment arms conducted at the Alfred Psychiatry Research Centre in Melbourne. Randomization will occur via the generation of a computer number sequence. Subjects will be randomized immediately prior to the commencement of the first treatment session, after the measurement of bilateral resting motor thresholds with standard means.

The main study phase (phase 1) will involve the 4 week randomized controlled trial conducted under strict double-blind conditions. Fidelity of the blinding process will be assessed at the end of this period with patients and raters. Phase 2 will involve the provision of open label treatment to patients who received sham treatment and wish to receive 'active' rTMS.

Responders to active treatment from phase 1 or 2 (defined as a 50% reduction in MADRS scores persisting for 1 week following the end of acute treatment) will enter phase 3, a 6 month maintenance phase. During this time, a single rTMS treatment session will be provided every week for 2 months and then every 2 weeks for 4 months. Acute treatment for up to 4 weeks will be reinstated if there is a persistent (2 week) increase in MADRS score of >25%.

ELIGIBILITY:
Inclusion criteria:

1. Be aged 18-60 and have capacity to consent
2. Currently meet DSM-IV criteria for a diagnosis of major depressive disorder (expect for the exclusion of causality by a general medical condition referring to the TBI) and have the persistence of depressive symptoms for at least one month at sufficient severity to warrant the diagnosis.
3. Have experienced a closed head injury of mild to moderate severity (Glasgow coma scale score (GCS) of greater than 8), preceding their depression, and are at least 3 months post injury. The injury must not have involved specific direct damage to either frontal lobe.
4. Have a Montgomery Asberg Rating Scale Score of > 20 (moderate - severe depression). Including only a more severely ill group of subjects limits the placebo response rate.
5. Have had no increase or initiation of new antidepressant (or other psychoactive) therapy in the 4 weeks prior to enrolment.

Exclusion Criteria:

1. Patients who have an unstable medical condition, neurological disorder or any history of a seizure disorder or are currently pregnant or lactating.
2. Patients who have experienced clear structural damage to the left or right dorsolateral prefrontal cortex as documented on MRI scan
3. Have a current DSM IV diagnosis of alcohol or substance dependence disorder.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Depression Symptom Severity | 4 weeks

SECONDARY OUTCOMES:
Cognitive Tasks | 4 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Fitzgerald, MBBS, FRANZCP, PhD, Principal Investigator — Alfred Psychiatry Research Centre
Locations (1):
- Alfred Psychiatry Research Centre, Prahran, Victoria, Australia